CLINICAL TRIAL: NCT04853108
Title: Using Telemedicine, Remote Physiologic Monitoring, and Mobile Self-reported Symptom Surveys to Improve Care for COVID-19 Patients
Brief Title: Remote Monitoring of COVID-19 Positive Outpatients
Status: Terminated | Type: Observational
Why Stopped: The study terminated early due to end of funding.
Sponsor: Emory University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Blake Anderson, Assistant Professor, Emory University
Other Study IDs: STUDY00001408
Record Dates: First submitted 2021-04-19; First posted 2021-04-21 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: Telemedicine; Risk assessment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remote Monitoring of COVID-19: Patients with COVID-19 who completed acute clinical monitoring of at least 30 days from symptom onset or positive COVID-19 test.
  Interventions: Other: Remote Monitoring of COVID-19

INTERVENTIONS:
Other: Remote Monitoring of COVID-19 — Remote monitoring of acute COVID-19 illness included use of a Medtronic pulse oximeter, photoplethysmography (PPG), patient-reported symptoms data, static vital signs captured during the course of the clinical evaluation and various physiomarkers.

SUMMARY:
This study seeks to evaluate how secondary data retrieved from remote physiological monitoring performed during routine outpatient/at-home care periods can allow for the discovery of novel physiomarkers that predict acute deterioration or hospitalization among people testing positive for Coronavirus Disease 2019 (COVID-19).

DETAILED DESCRIPTION:
Most recent research publications and clinical trials have exclusively focused on the hospital and intensive care unit (ICU) care of COVID-19 patients. Few have focused on how to direct care delivered at home, where the majority of coronavirus infected will recover, and how and when to rescue those who are at immediate risk for poor outcomes. To standardize the home monitoring process and offer guidance in this uncharted territory, the researchers have created a method for outpatient management of COVID-19 patients and high suspicion influenza-like illness (ILI) for Emory University Hospital. This includes the newly implemented model of clinics including in-person ambulatory management in the Acute Respiratory Clinic (ARC), the Virtual Outpatient Management Clinic (VOMC), and the Emory COVID-19 Outpatient Remote Monitoring Registry (E-CORMR). Initial analysis of the management system, particularly in risk tier assignment, has shown that assigning risk tiers early can help to identify patients at risk for clinical deterioration. The researchers have also demonstrated symptom profiles and durations of the "typical" outpatient disease course. The E-CORMR was used to create a dashboard for improved management of these frequently complex patients. It was determined after its creation that it could also be used for research purposes to store data collected from physiologic parameters.

The goal of this study is to develop algorithms using secondary data abstracted from remote monitoring devices that were collected within the E-CORMR. The researchers propose to derive robust algorithms through the analysis of that data that identify a potential hospitalization. The findings will not only improve the management of patients with known or suspected COVID-19 but also provide information that allows early intervention on patients at risk of decompensation. This information can then be used by other healthcare systems to care for patients more safely at home, thus reducing the impact of COVID-19 on overburdened acute care settings and preventing poor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* identified to be positive for COVID-19 by Quantitative Reverse Transcription polymerase chain reaction (qRT-PCR)
* demonstrate symptoms of COVID-19
* symptom onset within 7 days
* completed 21 days of remote monitoring with a Medtronic remote pulse oximeter device

Exclusion Criteria:

* none

Ages: 25 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is obtained from patients admitted to the hospital or enrolled in the Emory COVID-19 Outpatient Remote Monitoring Registry (E-CORMR) by nursing triage for suspicion of COVID-19.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Identify Parameters Associated with Adverse Outcomes | Up to 2 months after creation of the registry
  The Emory COVID-19 outpatient remote monitoring registry (E-CORMR) will be used to identify physiologic parameters and symptom responses that are associated with adverse outcomes.

SECONDARY OUTCOMES:
Develop Algorithm for Deterioration | Up to 2 months after creation of the registry
  The E-CORMR database will be used to develop a robust clinical algorithm for deterioration among patients with COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Blake Anderson, MD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic, Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No